CLINICAL TRIAL: NCT07129837
Title: Serum Anti-PCOLCE as Novel Diagnostic Biomarker in Rheumatoid Arthritis With Emphasis on Seronegative Patients.
Acronym: Anti-pcolce/RA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Mariam Rezk Lyas Ibrahim, Principal investigator, Assiut University
Other Study IDs: Anti-pcolce in RA
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Seronegative; Elisa; Anti-pcolce; Biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Patients: Adult patients (≥18 years) diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria.
  Interventions: Diagnostic Test: Clinical evaluation, disease activity and disability scoring, and laboratory testing including RF, anti-CCP, and serum anti-PCOLCE antibody measurement by ELISA.
- Healthy Controls: Age- and sex-matched healthy individuals without rheumatoid arthritis or other autoimmune diseases.

INTERVENTIONS:
Diagnostic Test: Clinical evaluation, disease activity and disability scoring, and laboratory testing including RF, anti-CCP, and serum anti-PCOLCE antibody measurement by ELISA. — For rheumatoid arthritis (RA) patients: participants will undergo comprehensive clinical evaluation including demographic data, detailed history, musculoskeletal and systemic examination, assessment of disease activity using DAS-28 score, functional disability evaluation by modified Health Assessment Questionnaire (mHAQ), and laboratory investigations including CBC, ESR, CRP, rheumatoid factor (RF), anti-cyclic citrullinated peptide (anti-CCP) antibodies, and serum anti-procollagen C-endopeptidase enhancer (anti-PCOLCE) antibodies measured by ELISA.
  For healthy controls: participants will undergo comprehensive clinical evaluation including demographic data, detailed history, musculoskeletal and systemic examination, and laboratory testing limited to serum anti-PCOLCE antibodies measured by ELISA.
  Other Names: Serum anti citrullinated procollagen c endopeptidase enhancer anti-bodies.; Serum Anti-pcolce
  Groups: Rheumatoid Arthritis Patients

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease that primarily affects synovial joints, leading to pain, swelling, and progressive joint damage. Early diagnosis is critical to prevent irreversible disability. However, up to 30% of RA patients are seronegative for conventional markers such as rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) antibodies, creating a diagnostic challenge. This study aims to evaluate the diagnostic performance of serum anti-procollagen C-endopeptidase enhancer (anti-PCOLCE) antibodies in RA patients, with a particular focus on seronegative cases. We will conduct a case-control study involving RA patients and age- and sex-matched healthy controls. Clinical assessments, disease activity scoring, functional disability evaluation, and laboratory testing will be performed. The findings may provide evidence for anti-PCOLCE as a novel biomarker for improved RA diagnosis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an inflammatory disease that primarily affects synovial joints through an autoimmune mechanism. If not treated properly, the disease can lead to bone erosion, joint deformities, and disability. Arthritis can also cause serious extra-articular disorders, including interstitial lung disease, vasculitis, and lymphoma.

The global prevalence of RA is 1%, with 44% of patients incapacitated within ten years. Increasing evidence indicates that early diagnosis and treatment of RA are crucial in preventing or delaying progression to erosive disease.

The production of antibodies to modified self-antigens is a hallmark in RA damage to synovial joints. The diagnosis of RA is based on a combination of clinical, radiographic, and serological findings. Among serological biomarkers, the most widely used are rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) antibodies. While anti-CCP antibodies are relatively specific for RA and are included in the 2010 ACR/EULAR classification criteria, they are not present in all patients. Approximately 20-30% of RA patients may test negative for both RF and anti-CCP, is termed seronegative RA (SNRA) emphasizing the need for additional, more sensitive and specific biomarkers, especially in early and seronegative RA.

Antibodies to citrullinated and carbamylated proteins are of particular interest in RA because of their high prevalence, specificity, association with erosive disease, and appearance during the preclinical phase of RA. Citrullination is a physiological posttranslational modification (PTM) best known for its role in gene regulation and skin keratinization. During this process, arginine residues are converted to citrulline by the activity of the peptidylarginine deiminase (PAD) enzymes.

Procollagen C-protease enhancer protein (PCOLCE) is a secretory glycoprotein, which plays an important role in enhancing the activity of procollagen C-Protease and promoting the reconstruction of extracellular matrix.

PCOLCE essential for the maturation of collagen, particularly types I and II. These collagen types are major components of articular cartilage and connective tissues. In the inflammatory environment of RA, PCOLCE can undergo citrullination, potentially converting it into a novel autoantigen.

Emerging evidence suggests that PCOLCE may elicit an autoimmune response in RA patients. Detecting autoantibodies directed against PCOLCE (anti- PCOLCE ) could therefore provide a new serological tool for RA diagnosis. These antibodies may not only enhance diagnostic accuracy particularly in patients who are seronegative for conventional markers but also shed light on novel mechanisms in RA pathophysiology.

ELIGIBILITY:
Inclusion criteria Adults (≥18 years old).

Patients clinically diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria:

Exclusion criteria Patients with other autoimmune or connective tissue diseases (e.g., SLE, SS). Patients with chronic infections or malignancies. Patients less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups will be included: rheumatoid arthritis patients attending the Rheumatology, Rehabilitation and Physical Medicine Department at Assiut University Hospital, and age- and sex-matched healthy controls recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Serum anti-PCOLCE antibody levels in rheumatoid arthritis patients versus healthy controls | Baseline (at the time of enrollment)
  To measure serum level of anticitrullinated procollagen C endopeptidase enhancer antibody (anti-PCOLCE) in RA patients compared to healthy controls .
  To assess the diagnostic performance of anti PCOLCE for RA specifically seronegative RA patients.
measure serum level of anticitrullinated procollagen C endopeptidase enhancer antibody (anti-PCOLCE) in RA patients compared to healthy controls . | At baseline (single measurement at enrollment).
  To measure serum level of anticitrullinated procollagen C endopeptidase enhancer antibody (anti-PCOLCE) in RA patients compared to healthy controls .
  To assess the diagnostic performance of anti PCOLCE for RA specifically seronegative RA.
  To evaluate correlation of serum anti-PCOLCE level with disease activity and functional disability scores in RA patients .

SECONDARY OUTCOMES:
Correlation between serum anti-PCOLCE antibody levels and disease activity scores in RA patients | At baseline (single assessment at enrollment).
  To assess the relationship between serum anti-procollagen C-endopeptidase enhancer (anti-PCOLCE) antibody levels and clinical disease activity and functional disability scores in RA patients , measured by DAS28-ESR, CDAI, and HAQ-DI scores.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Woude D, Young A, Jayakumar K, Mertens BJ, Toes RE, van der Heijde D, Huizinga TW, van der Helm-van Mil AH. Prevalence of and predictive factors for sustained disease-modifying antirheumatic drug-free remission in rheumatoid arthritis: results from two large early arthritis cohorts. Arthritis Rheum. 2009 Aug;60(8):2262-71. doi: 10.1002/art.24661. PMID 19644846
- [Background] Figus FA, Piga M, Azzolin I, McConnell R, Iagnocco A. Rheumatoid arthritis: Extra-articular manifestations and comorbidities. Autoimmun Rev. 2021 Apr;20(4):102776. doi: 10.1016/j.autrev.2021.102776. Epub 2021 Feb 17. PMID 33609792
- [Background] Maska L, Anderson J, Michaud K. Measures of functional status and quality of life in rheumatoid arthritis: Health Assessment Questionnaire Disability Index (HAQ), Modified Health Assessment Questionnaire (MHAQ), Multidimensional Health Assessment Questionnaire (MDHAQ), Health Assessment Questionnaire II (HAQ-II), Improved Health Assessment Questionnaire (Improved HAQ), and Rheumatoid Arthritis Quality of Life (RAQoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S4-13. doi: 10.1002/acr.20620. No abstract available. PMID 22588760
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27156434/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33609792/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22588760/